CLINICAL TRIAL: NCT01765933
Title: Pharmacokinetic and Physiological Effects of Oral DMAA Administration
Brief Title: Pharmacokinetic Effects of Oral DMAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: University of Tennessee (Other); USP Labs, Inc. (Industry)
Responsible Party: Principal Investigator, Brian Schilling, Associate Professor, University of Memphis
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DMAA Pharmacokinetics
Record Dates: First submitted 2013-01-08; First posted 2013-01-11 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Outcomes of Single Oral Dose
Keywords: 1,3-dimethylamylamine
MeSH Terms: interventions — 17-N,N-diethylcarbamoyl-4-methyl-4-azaandrostane-3-one; 1,3-dimethylamylamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DMAA (Experimental): Single oral dose 25 mg DMAA
  Interventions: Dietary Supplement: DMAA

INTERVENTIONS:
Dietary Supplement: DMAA — no placebo
  Other Names: 1,3-dimethylamylamine

SUMMARY:
1,3-dimethylamylamine (DMAA) has become increasingly popular as a component of dietary supplements. It is also used within "party pills," often in conjunction with alcohol and other drugs, and has been associated with untoward effects when abused at high dosages. To our knowledge, no studies have been conducted to determine the combined pharmacokinetic profile and physiologic responses of DMAA. To conclude on the safety profile of DMAA based solely on case reports would be problematic, in particular when accepting testimony from patients in uncontrolled environment, potentially under the influence of alcohol and other drugs. This is especially true in light of the fact that no prospective studies have shown these effects. Hence, the intent of the present study was to determine the pharmacokinetic profile of a single 25mg oral dosage of DMAA alone through 24 hours post-ingestion. This represents a typical dosage within one serving of many popular dietary supplements containing DMAA.

ELIGIBILITY:
Inclusion Criteria:

* must be able to swallow pill

Exclusion Criteria:

* self-reported cardiovascular or metabolic problems
* current smokers

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics | 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hr
  The area under the plasma concentration-time curve from time 0 to infinity was calculated using the trapezoidal rule extrapolated to time infinity. The terminal half-life (t 1/2) was calculated using 0.693/Lambda z, with Lambda z as the terminal rate elimination constant. Peak concentration (Cmax), lag time (tlag), time of maximum concentration (tmax), apparent volume of distribution during the terminal elimination phase (Vz/F), and oral clearance (CL/F) were also calculated.

SECONDARY OUTCOMES:
physiological effects on heart rate and blood pressure | 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hr
  heart rate, blood pressure

OTHER OUTCOMES:
cutaneous temperature | 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hr
  skin temperature

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Memphis, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Schilling BK, Hammond KG, Bloomer RJ, Presley CS, Yates CR. Physiological and pharmacokinetic effects of oral 1,3-dimethylamylamine administration in men. BMC Pharmacol Toxicol. 2013 Oct 4;14:52. doi: 10.1186/2050-6511-14-52. PMID 24090077